CLINICAL TRIAL: NCT07385716
Title: Evaluation of the Effect of Time-Restricted Feeding and Mediterranean Diet Model in Women With Polycystic Ovary Syndrome
Acronym: PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, SUHİDE BİLGE HORZUM, dietitian, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-12/51
Record Dates: First submitted 2026-01-17; First posted 2026-02-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Mediterranean diet; intermittent fasting
MeSH Terms: conditions — Polycystic Ovary Syndrome; Intermittent Fasting | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The study sample consists of women in Konya province who applied to the Healthy Living Center after a physician evaluation and were diagnosed with PCOS. To determine the number of participants, the GPower 3.1.9.7 power analysis program requires the inclusion of a total of 56 women, with at least 28 women in each group, using 80% power and a 0.05 margin of error (actual power = 0.8037085). Since the study is planned in a longitudinal-randomized controlled design, a total of 62 participants will be included, with 31 women in each group, taking into account a 10% dropout rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet group (Active Comparator): Mediterranean diet
  Interventions: Other: Mediterranean diet
- intermittent fasting group (Active Comparator): intermittent fasting
  Interventions: Other: intermittent fasting

INTERVENTIONS:
Other: Mediterranean diet — Participants following the Mediterranean diet model will be informed about the Mediterranean diet pyramid, and the dietitian will plan how often and in what portions olive oil, nuts, olives, fish, yogurt, fruits, and vegetables they should consume. The Mediterranean diet pyramid recommends the daily, weekly, and monthly consumption frequencies of these foods. Weekly, it recommends consuming fish and seafood at least twice a week, 2 portions of white meat, 2-4 portions of eggs, less than 2 portions of red meat, 1 portion or less of processed meat, and less than 3 portions of sweets. Daily, it recommends 2 portions of dairy products, 1-2 portions of olive oil-based seeds and nuts, and more spices, herbs, garlic, and onions. It is also emphasized that each main meal should include 1-2 portions of fruit, more than 2 portions of vegetables, and 1-2 portions of olive oil and whole grains. Portion sizes are adjusted to individual needs and will be supported by food r
  Arms: Mediterranean diet group
Other: intermittent fasting — The women with PCOS included in the study will be randomly divided into two groups: one following the Mediterranean diet model and the other the intermittent fasting diet model. In randomized controlled trials, it is desirable for the number of participants in each group to be equal, balanced, and share similar characteristics. In this way, each participant will be included in any group with an equal and known probability. In the study, the assignment of participants to the groups will be done using a simple randomization method and a randomizer program (https://www.random.org/). The time-restricted eating (TRF) model will be applied. The time restriction will be planned as an 8-hour eating and 16-hour fasting period, suitable for the individuals' lifestyles. For individuals who agree to participate in the study, the eating times will be set as 11:00-12:00 and 19:00-20:00. It will be stated that the group applying the TRF model can drink non-energy beverages such as water, tea, and min
  Arms: intermittent fasting group

SUMMARY:
Currently, there is still insufficient data to support the long-term efficacy, safety, and health benefits of time-restricted feeding models in women diagnosed with Polycystic ovary syndrome (PCOS), and further studies are needed to test and validate the effects of long-term dietary management in PCOS. On the other hand, similarly, studies investigating the effects of the Mediterranean Diet on body composition and dietary intake in women with PCOS are limited. The primary aim of this research is to examine the effect of time-restricted feeding and the Mediterranean diet model on body composition and dietary intake in adult women diagnosed with PCOS. The secondary aim is to evaluate the effect of different dietary models on quality of life in women diagnosed with PCOS.

DETAILED DESCRIPTION:
PCOS is the most common female endocrine disorder and is characterized by chronic anovulation, hyperandrogenism, and polycystic ovaries.

The term PCOS was first used in 1935 when menstrual irregularities, decreased fertility, obesity, and hirsutism were reported in patients. Amenorrhea and resulting infertility, obesity, and male-pattern hair growth were listed among the symptoms. Diagnosis was made in the 1970s and 1980s by measuring luteinizing hormone (LH) levels.

At a conference organized by the National Institute of Health in 1990, it was stated that the primary diagnostic criteria for PCOS are infrequent ovulation and symptoms of androgen excess. Since 2003, PCOS has been diagnosed when at least two of the three Rotterdam criteria are present. Clinical hyperandrogenism (with hirsutism, acne, seborrhea, and alopecia) and/or high circulating androgen levels, the presence of ovarian cysts assessed by ultrasound examination, and anovulation and/or oligo-amenorrhea are criteria that lead to diagnosis. Various interventions (pharmacological, non-pharmacological, or surgical) exist to reduce PCOS symptoms. Metformin is a commonly used insulin sensitizer in PCOS patients with insulin resistance, but gastrointestinal side effects limit its use as a first-line treatment for long-term management. The international evidence-based guidelines for the assessment and management of PCOS, updated in 2018, recommend diet and exercise therapies as the first step in management. These guidelines focus on improving diagnostic accuracy by significantly improving individual diagnostic criteria; The focus is on reducing unnecessary testing; increasing emphasis on education, lifestyle changes, emotional well-being and quality of life; and highlighting evidence-based medical treatment and cheaper and safer fertility management.

Diet and exercise interventions are important because 60% of women with PCOS are overweight or obese. Recently, various dietary interventions are being tried for the management of PCOS. Fasting is known as one of the oldest traditions in the world and is practiced among various communities for cultural or religious reasons. Fasting has also been used as a method of treating diseases in the past. Hippocrates, considered the father of modern medicine, emphasized the importance of fasting during illness with his words, "To eat when you are sick is to feed your sickness". Intermittent fasting (IF), that is, periods of voluntary abstinence from food and drink, is known as an ancient practice followed in different forms by many populations worldwide. With intermittent fasting, there is a state of fasting or restricted eating at certain times of the day or on certain days of the week. IF; It can be implemented in three different types: alternate-day fasting, 5:2 diet, and time-restricted eating (TRF). Alternate-day fasting involves alternating days when food and drinks are consumed with fasting days when energy-containing foods or drinks are not consumed. In alternate-day fasting, approximately 20-25% of the energy requirement is met on fasting days. Modified fasting diet is also known as the 5:2 method. In this nutritional model, 2 non-consecutive days of the week involve a very low-calorie diet, while the other 5 days include normal energy requirements without energy restriction. Another approach is time-restricted eating, which is used to describe an eating pattern where food intake is limited to a time window of 8 hours or less each day. Among intermittent fasting diets, the TRF diet is a lifestyle intervention that limits the duration of food intake to a fixed number of hours. Welton et al. reported that the ideal fasting duration for positive weight change is 16 hours. In recent years, small-scale human studies demonstrating the importance of time-restricted eating have become widespread. Most of these studies have revealed the beneficial aspects of intermittent fasting in human metabolism, as in animal studies. With TRF, reductions in energy intake, body weight, body fat, blood sugar, triglycerides, glucose tolerance, and inflammatory markers have been observed. It has been found that IF may be beneficial in reducing body weight, improving insulin resistance, and reducing infection by regulating the circadian rhythm, gut microbial composition, and metabolism. Disruption in the circadian rhythm; Because it is associated with insulin resistance, excessive androgen production, increased Anti-Müllerian Hormone (AMH) levels, and apoptosis of granulosa cells, TRF is predicted to alleviate PCOS by improving the circadian rhythm. In addition, IF diets can improve PCOS by reducing insulin resistance through the stimulation of AMP-activated protein kinase (AMPK). In a recent review, it was found that in overweight/obese women with PCOS, the 5:2 diet and TRF promised improvements in menstrual regulation by significantly reducing the free androgen index and increasing sex hormone binding globulin. In a study in which 30 women diagnosed with PCOS underwent a 6-week, 8-hour TRF diet intervention, baseline (pre-diet) and post-diet findings were compared. It was found that after the diet, body mass index (BMI) and body weight decreased significantly, HOMA-IR improved significantly, and metabolic parameters related to glucose and lipid profiles also showed significant improvements after the diet. The Mediterranean diet is considered a health-promoting dietary model due to its unique characteristics, including regular consumption of unsaturated fats, low glycemic index carbohydrates, high amounts of fiber, vitamins, antioxidants, and moderate amounts of animal-derived proteins. In addition to weight loss, it has been reported to have anti-inflammatory activity due to the production of short-chain fatty acids stimulated by dietary fiber. The Mediterranean diet pyramid recommends foods to be consumed daily, weekly, and monthly. It is recommended that fish and seafood be consumed at least twice a week, white meat in 2 servings, eggs in 2-4 servings, red meat in less than 2 servings, processed meat in 1 serving or less, and desserts in less than 3 servings. Daily, it is recommended that dairy products be consumed in 2 servings, and olive oil-based seeds and nuts in 1-2 servings.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-49 years of age
* Having been diagnosed with PCOS by a specialist according to Rotterdam criteria
* Having a BMI between 25-35 kg/m2
* Not having any conditions that impair reality testing and cognitive functions, preventing interviews or completing scales
* Being literature
* Having signed the informed consent form by agreeing to participate in the study.

Exclusion Criteria:

* Combination of other endocrine etiological disorders according to Rotterdam criteria (congenital adrenal hyperplasia, Cushing syndrome, androgen-secreting tumors, hyperprolactinemia, thyroid, adrenal and other endocrine disorders)
* Combination of cardiovascular and cerebrovascular diseases, hematological disorders, hepatic and renal failure and other serious diseases
* Liver and kidney disease
* Use of insulin or oral antidiabetic drugs,
* Being pregnant and lactating
* Low compliance and non-compliance with treatment during the intervention (individuals with less than 80% compliance will be excluded from the study)
* Preparation for pregnancy status during the dietary intervention
* Women with pacemakers or defibrillators implanted due to the theoretical possibility of interference with device activity due to the current field caused by impedance measurements
* Use of medication affecting carbohydrate or lipid metabolism in the last 6 months (oral contraceptive pills, insulin sensitizers, antiepileptics, antipsychotics, statins and fish oil)
* A psychiatric condition diagnosed by a physician It has been determined as a disease state.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Polycystic Ovary Syndrome Quality of Life-50 Scale (PCOSQ-50) | 8 weeks
  Consisting of 50 questions and 6 parameters, the scale's parameters are psychosocial and emotional status, fertility, sexual function, obesity and menstrual irregularity, hirsutism, and coping with the disease. The PCOSQ-50 scale is scored using a scale of always 1, frequently 2, sometimes 3, rarely 4, and never 5. Thus, the total score can range from 50 to 250 points. A lower score indicates a lower quality of life, while a higher score indicates less or no effect on quality of life. The Turkish validity and reliability study of the scale was conducted by Koyutürk (2018). The internal consistency coefficient (Cronbach's alpha) of the PCOSQ-50 scale is 0.972, and the internal consistency coefficients of the sub-dimensions range from 0.956 to 0.977. In this study, the Cronbach alpha value is 0.936.

SECONDARY OUTCOMES:
Body fat percentage (% fat) | 8 weeks
  Individuals' body weights and body compositions will be measured using foot-to-foot bioelectrical impedance analysis (BIA). Body fat percentage (% fat) will be measured using a TANITA MC 580.
Body mass index (BMI) | 8 weeks
  Body mass index (BMI) will be calculated using the equation where body weight is divided by the square of height in meters, and will be evaluated according to the World Health Organization's classification for adults.
blood glucose (mg/dL) | 8 weeks
  All participants included in the study will be informed that they can return to their primary care physician at the end of the 8th week for an evaluation of their medical nutrition therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province have routine biochemical tests performed at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. Fasting blood glucose (mg/dL) values of individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
weight | 8 weeks
  Individuals' body weights and body compositions will be measured using foot-to-foot bioelectrical impedance analysis (BIA). Weight will be measured in kilograms and the measurement will be performed using a TANITA MC 580 device.
Serum insulin (μIU/mL) | 8 weeks
  All participants included in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutrition therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province have routine biochemical tests performed at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. Serum insulin (μIU/mL) values of individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
HbA1C (%) | 8 weeks
  All participants in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutrition therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province perform routine biochemical tests at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of basic health care will be used as data. The HbA1C (%) values of the individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
Total Cholesterol (mg/dL) | 8 weeks
  All participants included in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutritional therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province perform routine biochemical tests at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. Total Cholesterol (mg/dL) values of individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
LDL (mg/dL) | 8 weeks
  All participants included in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutrition therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province perform routine biochemical tests at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. LDL (mg/dL) values of individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
HDL (mg/dL) | 8 weeks
  All participants included in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutrition therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province perform routine biochemical tests at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. The HDL (mg/dL) values of the individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.
Triglyceride (mg/dL) | 8 weeks
  All participants included in the study will be informed that they can revisit their primary care physician at the end of the 8th week for an evaluation of their medical nutritional therapy, and their biochemical findings will be recorded on the research form. Since all primary care physicians in the same province perform routine biochemical tests at the same reference laboratory, all results obtained retrospectively from patients are standardized. No invasive procedures will be performed specifically for this research. No biochemical tests specific to this study will be conducted; only the results of routine biochemical tests already performed within the scope of patients' basic health care will be used as data. Triglyceride (mg/dL) values of individuals participating in the study will be recorded retrospectively on the data collection form before the diet and after the 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Melda Kangalgil, Principal Investigator — Cumhuriyet University; Ayşe N Kahve, Principal Investigator — Aksaray University
Locations (1):
- Healthy Life Center, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Polycystic Ovary Syndrome Quality of Life-50 Scale (PCOSQ-50) Biochemical Parameters Anthropometric Measurements
Supporting Information: Study Protocol, ICF
Time Frame: January 2026 - March 2026
Access Criteria: The aim is to benefit society by publishing the study results at the end of the study.

REFERENCES:
- [Result] Barrea, L., Arnone, A., Annunziata, G., Muscogiuri, G., Laudisio, D., Salzano, C., Pugliese, G., Colao, A., & Savastano, S. (2019). Adherence to the Mediterranean diet, dietary patterns and body composition in women with polycystic ovary syndrome (PCOS). Nutrients, 11(10), 2278